CLINICAL TRIAL: NCT04175327
Title: Post-Market Registry in Europe for the Use of CardioCel®, CardioCel® Neo and CardioCel® 3D
Brief Title: Prospective and Non-randomized Registry of CardioCel 3D
Status: Active, not recruiting | Type: Observational
Sponsor: LeMaitre Vascular (Industry)
Collaborators: Factory CRO for Medical Devices B.V. (Other)
Responsible Party: Sponsor
Other Study IDs: GLRA-G010
Record Dates: First submitted 2019-11-19; First posted 2019-11-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Intracardiac and Septal Defects; Valve and Anulus Repair; Great Vessel Reconstruction; Peripheral Vessel Reconstruction; Suture Line Buttressing
MeSH Terms: conditions — Heart Septal Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CardioCel group: Patients who require repair of cardiac and vascular defects including intracardiac defects; septal defects, valve and annulus repair; great vessel reconstruction, peripheral vascular reconstruction and suture line buttressing
  Interventions: Device: CardioCel implantation

INTERVENTIONS:
Device: CardioCel implantation — treatment of intracardiac defects; treatment of septal defects; valve and annulus repair; great vessel reconstruction; peripheral vascular reconstruction; suture line buttressing

SUMMARY:
Post-market, prospective, multi-centre, open-label, registry designed to collect prospective safety and performance data on the use of CardioCel in patients with cardiovascular disorders and in accordance with local standard of care.

The Registry will collect data with a minimum of 50 subjects per major indication (minimum total of 200) in 5-10 sites in Europe. The clinical investigation will maintain data for each patient from the date of implant through 2 years post-implantation.

DETAILED DESCRIPTION:
Post-market, prospective, multi-centre, open-label, registry designed to collect prospective safety and performance data on the use of CardioCel in patients with cardiovascular disorders and in accordance with local standard of care. The Registry has been designed to collect prospective product safety and performance data after the CardioCel line extension for CardioCel 3D and the indication expansion to include great vessel and peripheral reconstruction and suture line buttressing and will collect safety and performance data up to 2 years following implantation. The CardioCel 3D Registry will collect data on the use of the CardioCel,

CardioCel Neo and CardioCel 3D for the following major indications:

* Intracardiac and septal defects
* Valve and annulus repair
* Great vessel reconstruction
* Peripheral vascular reconstruction

As suture line buttressing is a procedure that does not consistently use tissue, data on this indication will only be included if available. Data will be prospectively collected by the sites on registry-specific electronic case report forms (eCRFs). The primary endpoints will assess devices' safety and performance through measures and images obtained via the facility's standard of care at the respective registry site. Additional data will also be collected from the implant procedure to assess user (surgeon) satisfaction with the devices' handling and performance.

ELIGIBILITY:
Inclusion Criteria:

* patient has signed the informed consent
* patient is a candidate for treatment with CardioCel/CardioCel Neo/CardioCel 3D per approved device indications.

Exclusion Criteria:

- no study specific exclusion criteria; patients treated per standard clinical practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CardioCel, CardioCel Neo and CardioCel 3D are indicated for the repair of cardiac and vascular defects including intracardiac defects; septal defects, valve and annulus repair; great vessel reconstruction, peripheral vascular reconstruction and suture line buttressing.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of graft related reintervention | 30 days post procedure.
  capture the rate of graft related reintervention
Incidence of patch related morbidity | 30 days post procedure
  capture the rate of patch related morbidity

SECONDARY OUTCOMES:
Incidence of graft related reinterventions | at 1 and 2 years post-procedure
  capture the rate of graft related reinterventions
Rates of Valvular Regurgitation Grade > Moderate | 30 days post procedure
  for Valve and annulus repair
Rates of re-stenosis | at 30 days and 1 and 2 years follow-up
  for Great vessel reconstruction
Rates of recoarctation | at 30 days and 1 and 2 years follow-up
  for Great vessel reconstruction
Rates of measurement of the dynamic flow by facility standard of care ≥110-175* cm/sec for peripheral vascular locations | at 30 days and 1 and 2 years follow-up
  for Peripheral vascular reconstruction
incidence of Patch dehiscence | at 30 days and 1 and 2 years follow-up
  capturing the rate of patch dehiscence
Incidence of Patch calcification | at 30 days and 1 and 2 years follow-up
  capturing the rate of patch calcification
Incidence of Patch retraction | at 30 days and 1 and 2 years follow-up
  capturing the rate of patch retraction
Incidence of Unanticipated events | at 30 days and 1 and 2 years follow-up
  capturing the rate of unanticipated events

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Ghiu, Study Director — Anteris
Locations (6):
- Heart Center Leipzig, Leipzig, Germany
- Italy (2):
  - Policlinico San Donato, San Donato Milanese, MI
  - A.O.U. Città della Salute e della Scienza, Turin
- Hospital Universitario "Doce de Octubre", Madrid, Spain
- United Kingdom (2):
  - Bristol Children's Hospital and the Heart Institute, Bristol
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No